CLINICAL TRIAL: NCT01788852
Title: Prevalence of HPV and Intraepithelial Neoplasia Biomarkers in Adolescents
Brief Title: HPV in Adolescents
Status: Completed | Type: Observational
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Thai Red Cross AIDS Research Centre (Other); Chulalongkorn University (Other); SEARCH Research Foundation (Other); We Understand Group (Unknown); TREAT Asia (Unknown)
Responsible Party: Sponsor
Other Study IDs: HIV-NAT 139
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: HPV Infection; Cervical/Anal Dysplasia
Keywords: HPV; HIV; cervical/anal dysplasia; intraepithelial neoplasia; E6/E7 biomarker; perinatally HIV-infected adolescents; behaviorally HIV-infected adolescents; anal and pap smear
MeSH Terms: conditions — Papillomavirus Infections; Carcinoma in Situ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cervical and anal pap smears specimens will be used for HPV typing. Blood will be collected for STI and immune response to HPV/HIV testing
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Perinatally HIV-infected adolescents: Perinatally HIV-infected adolescents
- behaviorally HIV-infected adolescents: behaviorally HIV-infected adolescents
- HIV negative adolescents: HIV negative adolescents

SUMMARY:
This study will assess the prevalence of HPV infection in perinatally HIV-infected adolescents, intraepithelial neoplasia, and E6E7 biomarker at cervical and anal sites.

DETAILED DESCRIPTION:
Human Papillomavirus (HPV) is the most common sexually transmitted disease and it causes cervical and anal cancer. Prevalence and incidence of HPV infection among young adults who are sexually experienced is high. No data exist for HIV-positive adolescents in regards to HPV infection, cervical and anal intraepithelial neoplasia. This study will compare the prevalence of HPV infection, intraepithelial neoplasia and E6/E7 biomarker at cervical and anal sites among perinatally HIV-infected adolescents, behaviorally HIV-infected adolescents, and HIV-negative adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Perinatally-infected (documented positive HIV enzyme immunoassay (EIA) or nucleic acid testing (NAT) at any time and history of maternal HIV infection)
* behaviorally-infected (documented positive HIV enzyme immunoassay (EIA) or nucleic acid testing (NAT) at any time after sexual debut without history of maternal HIV infection)
* female with vaginal or receptive anal intercourse with a male OR male with receptive rectal intercourse with another male
* Signed informed consent. Volunteers aged 12-17 years can decide whether they wish for their parents to consent for their participation. Due to the confidential nature of the issues being studied, parental consent may be exempted

Exclusion Criteria:

* Have any conditions that may interfer with subjects' ability to understand and consent to the study

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A total of 60 sexually active adolescents (perinatally and behaviorally HIV-infected adolescents, HIV negative adolescents) aged 12-24 will be recruited from the HIV-NAT and TRC Anonymous Clinic
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
HPV infection | 48 weeks
  Prevalence of cervical and anal HPV infection and of oncogenic subtypes, among perinatally HIV-infected adolescents, behaviorally HIV-infected adolescents, and HIv-negative adolescents

SECONDARY OUTCOMES:
intraepithelial neoplasia | 48 weeks
  Prevalence of intraepithelial neoplasia among the three study groups and in male and female subjects
E6/E7 | 48 weeks
  Prevalence of detected E6/E7 biomarker among the tree study groups and in male and female subjects.
  Correlation between detected E6/E7 and presence of HPV infection and/or intraepithelial neoplasia Association between HAART use, CD4 counts, plasma HIV RNA level and HIV clinical staging with HPV infection, intraepithelial neoplasia and E6/E7 detection
HPV vaccine | 48 weeks
  Proportion of adolescents who would benefit from the current preventive vaccine (i.e. those who have not been infected with oncogenic HPV subtypes 16 and 18)

CONTACTS AND LOCATIONS:
Overall Officials: Jintanat Ananworanich, MD, PhD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration; Nittaya Phanuphak, MD, Principal Investigator — Thai Red Cross AIDS Research Centre
Locations (3):
- Thailand (3):
  - Department of Pediatrics, Chulalongkorn University, Bangkok
  - HIV-NAT, Bangkok
  - Thai Red Cross - Anonymous Clinc, Bangkok

REFERENCES:
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT)'s website — http://www.hivnat.org